CLINICAL TRIAL: NCT00738556
Title: Spot Drug-Eluting vs Full Cover Stenting for Long Coronary Stenoses: a Randomized Clinical Study
Brief Title: Spot Drug-Eluting Stenting for Long Coronary Stenoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiovascular Research Society, Greece (Other)
Responsible Party: Department of Cardiology, Athens Euroclinic
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2.15.8.08
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Angioplasty
MeSH Terms: interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Full cover stenting of coronary lesions
  Interventions: Device: Drug-eluting stents (Cypher and Taxus)
- 2 (Active Comparator): Spot-stenting of significantly stenotic parts of a coronary lesion
  Interventions: Device: Drug-eluting stents (Cypher and Taxus)

INTERVENTIONS:
Device: Drug-eluting stents (Cypher and Taxus) — Spot or full length stenting of a coronary lesion
  Other Names: Sirolimus-eluting stents (Cypher, J&J); Paclitaxel-eluting stents (Taxus, Boston Scientific)

SUMMARY:
Most doctors who use the new drug-eluting stents for the treatment of long coronary narrowings tend to cover the full length of the lesion with long or multiple stents. The investigators hypothesized that a policy of spot-stenting, i.e., stenting of only the very tight parts of the coronary narrowing, might result in better outcomes by means of avoiding multiple stents that have been associated with significant complications such as late stent thrombosis.

DETAILED DESCRIPTION:
Coronary artery lesion length is an independent predictor of restenosis following coronary intervention and the deployment of multiple or long bare metal stents has been associated with an increased risk of adverse clinical outcome. Spot stenting, ie discrete stenting of only the most severe stenoses of long, diffuse lesions has been proposed as an alternative in this clinical setting. The introduction of drug-eluting stents has resulted in longer lesions being stented and the use of multiple, overlapping DES in patients with diffusely diseased coronary arteries has been considered safe and effective. However, there has also been evidence of increased major adverse cardiac events (MACE) with the use of multiple, overlapping DES,10-12 while long DES have been associated with increased probability of intraprocedural stent thrombosis.13 We hypothesized that an approach based on spot-stenting with the use of DES might result in superior clinical outcomes compared to full cover of atheromatic lesions with long or multiple stents. We are therefore conducting a randomized comparison of spot versus multiple overlapping stenting on consecutive patients with long (>20 mm) lesions and indications for percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Consenting, consecutive patients with a de novo, native coronary artery lesion longer than 20 mm.

Exclusion Criteria:

* Unprotected left main coronary artery stenosis,
* Left ventricular ejection fraction <25%, OR
* Contraindication to aspirin or clopidogrel

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2003-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Demosthenes Katritsis, MD, PhD, Study Chair — Athens Euroclinic and Cardiovasdcular Research Society
Locations (2):
- Greece (2):
  - Athens Euroclinic, Athens, Attica
  - Athens Euroclinic, Athens

REFERENCES:
- [Background] Katritsis DG, Korovesis S, Karabinos I, Giazitzoglou E, Theodorou S, Karvouni E, Voridis E. Sirolimus-versus paclitaxel-eluting stents: a comparison of two consecutive series in routine clinical practice. J Interv Cardiol. 2006 Feb;19(1):31-7. doi: 10.1111/j.1540-8183.2006.00101.x. PMID 16483337
- [Background] Katritsis DG, Korovesis S, Karvouni E, Giazitzoglou E, Theodorou S, Kourlaba G, Panagiotakos D, Voridis E. Direct versus predilatation drug-eluting stenting: a randomized clinical trial. J Invasive Cardiol. 2006 Oct;18(10):475-9. PMID 17235419
- [Background] Karvouni E, Korovesis S, Katritsis DG. Very late thrombosis after implantation of sirolimus eluting stent. Heart. 2005 Jun;91(6):e45. doi: 10.1136/hrt.2004.056341. PMID 15894746
- [Background] Katritsis DG, Karvouni E, Ioannidis JP. Meta-analysis comparing drug-eluting stents with bare metal stents. Am J Cardiol. 2005 Mar 1;95(5):640-3. doi: 10.1016/j.amjcard.2004.10.041. PMID 15721109